CLINICAL TRIAL: NCT06108167
Title: Percutaneous Imaging-guided Cryoblation of the Anterior Abdominal Wall Endometriosis Scars
Acronym: ENDOMET
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8955
Record Dates: First submitted 2023-08-28; First posted 2023-10-30 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-08

CONDITIONS: Endometriosis
Keywords: Endometriosis; Endometrial cells; Radiofrequency; Anterior abdominal; Cryotherapy
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Endometriosis is a common condition affecting 10% of women. It is characterized by the presence of ectopic endometrial cells. This pathology most frequently develops in the ovaries, utero-sacral ligaments and pelvic peritoneum, but also in the recto-sigmoid. Rarely, these lesions are found outside the pelvis, and even more exceptionally in the abdominal wall (in 0.03 to 1% of cases).

Cryotherapy has already been used for many years to treat soft tissue tumors (kidney and prostate tumors). It has also been successfully used by interventional radiologists to treat parietal desmoid tumors. After discussions with radiologists, given the similarity of location and extension of wall endometriosis lesions with desmoid tumours, the successes observed, and the scarcity of studies in the literature, it seemed appropriate to the investigators to study this new therapy.

The aim of this study was to investigate the efficacy of cryotherapy on parietal endometriosis lesions.

ELIGIBILITY:
Inclusion Criteria:

* Adult woman (≥18 years old) Having benefited from cryotherapy of an abdominal wall endometriosis nodule between January 6, 2020 and January 2, 2023.
* Subject not objecting to the reuse of their data for the purposes of this research

Exclusion Criteria:

* Subject having expressed its opposition to the reuse of its data for scientific research purposes.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult woman (≥18 years old) Having benefited from cryotherapy of an abdominal wall endometriosis nodule between January 6, 2020 and January 2, 2023.
Sampling Method: Non-Probability Sample
Enrollment: 29 (Estimated)
Dates: Start 2023-05-05 (Actual); Primary Completion 2023-11-05 (Estimated); Study Completion 2023-11-05 (Estimated)

PRIMARY OUTCOMES:
Efficacy of cryotherapy on parietal endometriosis lesions was assessed using the a visual analogue scale (VAS) ranging from 0 to 10. | Before and 6 months after the cryotherapy

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Gynécologie Obstétrique - CHU de Strasbourg - France, Strasbourg, France